CLINICAL TRIAL: NCT05895032
Title: Development Of a haemophiLia PHysiotherapy INtervention for Optimum Musculoskeletal Health in Children (DOLPHIN-II) - a Randomised Controlled Trial
Brief Title: Trial of an Exercise Intervention for Children With Haemophilia
Acronym: DOLPHIN-II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: East Kent Hospitals University NHS Foundation Trust (Other Government)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other); University of Kent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020/HAEMO/01
Record Dates: First submitted 2020-07-21; First posted 2023-06-08 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Hemophilia; Child, Only; Musculoskeletal Diseases or Conditions
Keywords: Physical Therapy; Exercise; Muscle strength
MeSH Terms: conditions — Hemophilia A; Musculoskeletal Diseases; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A single-blinded, two-arm pragmatic randomised controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: It is impossible to blind those in receipt and those delivering the intervention as to group allocation. However, it will be possible, although perhaps challenging, to blind the assessor to group allocation. Consequently, we will attempt a single blind approach in which the participant and physiotherapists delivering the intervention will be encouraged to withhold their group allocation from the assessors collecting data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): 12-week exercise intervention
  Interventions: Other: Exercise
- Usual care (Active Comparator): Participants will continue to receive their usual care as prescribed by the haematologist, physiotherapist and other members of the healthcare team.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Exercise — 12-week exercise intervention
  Arms: Exercise
Other: Usual Care — usual care
  Arms: Usual care

SUMMARY:
"Being able to participate in games and activities with their friends" is one of the things that matters most to boys with haemophilia. At present, there is a lack of robust evidence to determine whether muscle strengthening exercise can improve or negatively affect outcomes for young children with haemophilia. With the help of boys with haemophilia, their parents and physiotherapists the investigators have developed an exercise programme designed to increase muscle strength. Using this intervention the investigators will undertake a single-blinded, two-arm pragmatic randomised controlled trial (RCT) of a 12-week intervention verses usual care of boys with haemophilia aged 6-12 years of age.

DETAILED DESCRIPTION:
Children are born with haemophilia. Females carry the disorder and usually males are affected. It is a disorder affecting 1:10000 people where the blood does not clot normally, leading to bleeding into muscles and joints. As a result, muscles become weak. Joints become painful and difficult to move. "Being able to participate in games and activities with their friends" is one of the things that matters most to boys with haemophilia. "What is the role of exercise for both prevention and treatment of joint damage in haemophilia?" is one of the top unanswered questions that concern patients, carers and healthcare professionals most. At present, there is a lack of robust evidence to determine whether muscle strengthening exercise can improve or negatively affect outcomes for young children with haemophilia. With the help of boys with haemophilia, their parents and physiotherapists the investigators have developed an exercise programme designed to increase muscle strength. The investigators think the exercise programme might have an effect on pain and movement in participants joints, help them participate in games and activities with their friends and improve their health in the long term. The investigators recently showed the exercise programme had no harmful effects, was acceptable to children with haemophilia and that the participants were willing to participate in a study to answer the question, "does muscle strengthening help improve the long term health of children with haemophilia?" To answer this question, the investigators will allocate 66 boys with haemophilia to a group that is asked to complete the 12-week exercise routine to strengthen their leg muscles and another 66 boys to a group that does not do the exercises. The boys will be allocated at random, so that each boy has an equal chance of being in either group. Random allocation helps ensure that two similar groups of boys will be compared. The investigators will monitor the boys throughout the study by measuring their muscle strength, how far they can walk in six-minutes and time taken to ascend and descend 12 steps. The investigators will also record how physically active the boys are using a wrist band as well as how satisfied they are with their health. The study will be managed by a group of health care professionals and researchers with experience and expertise in carrying out this type of research. In addition, the investigators will include parents of boys with haemophilia in the research team to provide invaluable lived experience of living with the condition. So that people hear about what the investigators learn in the study, the investigators will report the findings to other researchers using journals, relevant health care professionals through face to face meetings, and children with haemophilia and their families through newsletters and presentations at Haemophilia Society meetings.

ELIGIBILITY:
Inclusion Criteria:

• Children aged 6-12 years, with severe or moderate haemophilia A or B

Exclusion Criteria:

* von Willebrand disease
* past history of fracture or trauma to the lower limb
* orthopaedic surgery
* acquired brain injury or any other disturbance of the central nervous system; joint or muscle bleed in the lower limb in the past 6 weeks
* presence of lower limb pain or unable to fully comply with verbal instructions.

Ages: 6 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 132 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Muscle strength of the dominant knee extensors at 24 weeks | 24-weeks
  Maximum isometric torque (Newton.metres/kilogram of body weight)

SECONDARY OUTCOMES:
Muscle strength of the ankle plantarflexors and non-dominant knee extensors at 24 weeks | 24 weeks
  maximum isometric torque (Newton.metres/kilogram of body weight)
Bleeding episodes and coagulation factor usage | 24 weeks
  Number of bleeding episodes (number) and amount of coagulation factor used for treatment (number)
Six-minute timed walk (6MTW) | 24 weeks
  Distance walked in 6 minutes (metres)
Timed up and down stairs (TUDS) | 24 weeks
  Time taken to ascend and descend a flight of 12 steps (seconds)
Participation in physical activity | 24 weeks
  Time spent in moderate-vigorous physical activity physical activity (MVPA)
Child Health Utility 9D (CHU9D) | 24 weeks
  a paediatric preference based measure of health related quality of life (utility values on the 0.0 to 1.0 quality adjusted life year scale) Higher score represent higher adjusted life years.

CONTACTS AND LOCATIONS:
Overall Officials: David Stephensen, PhD, Study Chair — East Kent Hospitals University NHS Foundation Trust
Locations (1):
- Haemophilia Centre, Canterbury, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We do not have consent to share individual participant data